CLINICAL TRIAL: NCT03415074
Title: Ketoanalogue-supplemented Low Protein Diet and Deferring Dialysis in Patients With Severe Proteinuria and Advanced Diabetic Kidney Disease
Brief Title: Could Ketoanalogue-supplemented Low Protein Diet Defer Dialysis in Advanced Diabetic Kidney Disease? (K-DDD)
Acronym: K-DDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anemia Working Group Romania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AnemiaWGRomania
Record Dates: First submitted 2017-12-30; First posted 2018-01-30 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: CKD Stage 4
Keywords: low protein diet; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Intervention Model Description: Eligible patients will enter a run-in phase (3 mo), when mild protein diet (0.8g/kg dry ideal bw) will be initiated and compliance will be evaluated twice monthly.
  Those who will prove compliant during the run-in phase and still fulfill the selection criteria will be randomized 1:1 (computer-generated numbers) to receive the low protein diet (0.6 g/kg-day, mainly vegetarian) supplemented with ketoanalogues of essential amino-acids (Ketosteril 1 tb/10 kg dry bw) or to continue the mild protein restriction (0.8 g/kg-day).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemented low protein diet (sLPD) (Active Comparator): Protein restriction to a low level (0.6 g/kg-day, mainly vegetarian) + ketoanalogues of essential amino-acids supplementation (Ketosteril 1 tb/10 kg dry bw)
  Interventions: Behavioral: Protein restriction
- Mild protein restriction diet (MPD) (Active Comparator): Mild restriction in dietary protein intake (0.8 g/kg-day)
  Interventions: Behavioral: Protein restriction

INTERVENTIONS:
Behavioral: Protein restriction — In both arms the dietary protein intake will be reduced. In the sLPD arm, the protein restriction is more severe and ketoanalogues of the essential aminoacids are offered.

SUMMARY:
This is a prospective single center open label randomized controlled trial aiming to assess the effectiveness and safety of a low protein diet (0.6 g/kg-day, mainly vegetarian) supplemented with ketoanalogues of essential amino-acids (sLPD) as compared to a mild protein restriction (0.8 g/kg-day, MPD) in reducing Chronic Kidney Disease (CKD) progression, with a planned total duration is of 18 months.

Adult diabetic patients with CKD stage 4+ [estimated glomerular filtration rate (eGFR) using the Modification of Diet in Renal Disease 4-variable (MDRD4) formula <30 mL/min per year], with stable renal function (historical reduction of eGFR of < 10 ml/min-year) , proteinuria > 3g/g creatininuria and good nutritional status (SGA A) will be enrolled.

DETAILED DESCRIPTION:
Adult diabetic patients with Chronic Kidney Disease (CKD) stage 4+ (estimated GFR using the Modification of Diet in Renal Disease 4-variable, MDRD4, formula <30 mL/min per year), with stable renal function (historical reduction of eGFR of < 10 ml/min-year), proteinuria > 3g/g creatininuria and good nutritional status (SGA A) will be enrolled. Patients with evidence of active kidney disease (except proteinuria), with indication of etiological or pathogenic treatment, those with poor control of diabetes (HbA1c >8%), those with uncontrolled high blood pressure (≥155/85 mmHg), those with significant co-morbidities (heart failure, active liver disease, malabsorption, active infections, inflammatory diseases requiring corticosteroids), those with uremic symptoms (pericarditis, digestive disorders ) or malnutrition (SGA B or C, serum albumin < 3.5 g/dl) will be excluded.

Eligible patients will enter a run-in phase (3 mo), when mild protein restriction (0.8g/kg dry ideal bw) will be initiated and compliance will be evaluated twice monthly.

Those who will prove compliant during the run-in phase and still fulfill the selection criteria will be randomized 1:1 (computer-generated numbers) to receive the low protein diet (0.6 g/kg-day, mainly vegetarian) supplemented with ketoanalogues of essential amino-acids (Ketosteril 1 tb/10 kg dry bw) or to continue the mild protein restriction (0.8 g/kg-day).

The total recommended energy intake is of 30 kcal/kg of ideal dry body weight per day in all patients.

The primary composite endpoint is the need for RRT initiation or a more than 50% reduction in the initial eGFR any time during the assessment phase. The decision to initiate RRT will be made by the Ethical Committee of the Hospital, based on the clinical and laboratory data.

The need for RRT initiation, the quality of life [assessed by the Short Form-36 (SF-36) Questionnaire], the decline in GFR and the correction of metabolic complications of CKD [serum levels of urea, calcium, phosphates, serum parathyroid hormone levels, bicarbonate, potassium] will be secondary efficacy parameters.

Parameters of nutritional status (SGA, anthropometric and biochemical parameters), compliance to the diet, occurrence of any adverse event and the number of withdrawals will be safety variables.

All the parameters will be assessed at baseline, throughout the intervention phase and at end of the study.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients
* CKD stage 4+ (estimated GFR using the Modification of Diet in Renal Disease 4-variable, MDRD4, formula <30 mL/min per year)
* stable renal function (historical reduction of eGFR of < 10 ml/min-year)
* proteinuria > 3g/g creatininuria
* good nutritional status (SGA A)

Exclusion Criteria:

* evidence of active kidney disease (except proteinuria)
* indication for etiological or pathogenic treatment
* poor control of diabetes (HbA1c >8%)
* uncontrolled high blood pressure (≥155/85 mmHg)
* significant co-morbidities (heart failure, active liver disease, malabsorption, active infections, inflammatory diseases requiring corticosteroids)
* uremic symptoms (pericarditis, digestive disorders
* or malnutrition (SGA B or C, serum albumin < 3.5 g/dl)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
CKD progression | 15 months
  Percentage of patients requiring RRT initiation or a more than 50% reduction in the initial eGFR at anytime during the study

SECONDARY OUTCOMES:
Need for renal replacement therapy (RRT) | 15 months
  Percentage of patients requiring RRT during the study
Patients' Quality of life | at baseline and than every 3 months up to 15 months
  Patients' Quality of life, assessed by the SF-36 Questionnaire
Decline in eGFR | monthly up to 15 months
  Difference between eGFR at any timepoint and the initial eGFR
Correction of nitrogen balance | monthly up to 15 months
  Serum urea
Correction of metabolic acidosis | monthly up to 15 months
  Serum bicarbonate
Correction of calcium metabolism abnormalities | monthly up to 15 months
  Serum calcium
Correction of mineral metabolism abnormalities | monthly up to 15 months
  Serum phosphates
Serum level of intact Parathyroid Hormone (iPTH) | monthly up to 15 months
  iPTH
Nutritional status - Subjective Global Assessment (SGA) | monthly up to 15 months
  SGA
Body Mass Index (BMI) | monthly up to 15 months
  BMI
Tricipital Skin Fold (TSF) | monthly up to 15 months
  TSF
Middle arm muscular circumference (MAMC) | monthly up to 15 months
  MAMC
Serum albumin | monthly up to 15 months
  Serum albumin
Serum cholesterol | monthly up to 15 months
  Serum cholesterol
Inflammatory status | monthly up to 15 months
  Serum C-Reactive Protein (CRP)
Compliance to the protein intake | twice-a-month during the run-in phase, weekly for the first month after randomization, every 4 weeks during the next 6 months, and then every 3 months up to 15 months
  Achieved protein intake (urinary urea excretion, Mitch-Maroni's formula)
Compliance to the energy intake | twice-a-month during the run-in phase, weekly for the first month after randomization, every 4 weeks during the next 6 months, and then every 3 months up to 15 months
  Achieved energy intake (3-days food dairy)
Occurence of the adverse events | twice-a-month during the run-in phase, weekly for the first month after randomization, every 4 weeks during the next 6 months, and every 3 months up to 15 months
  Occurence of any adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mircescu, Prof, Study Chair — Carol Davila University of Medicine and Pharmacy
Locations (1):
- "Dr Carol Davila" Teaching Hospital of Nephrology, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
Unique patient number in the study, biological data; no data to enable patient identification will be provided
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: March 2022

REFERENCES:
- [Derived] Mihalache A, Garneata L, Mocanu CA, Simionescu TP, Mircescu G. Low-salt low-protein diet and blood pressure control in patients with advanced diabetic kidney disease and heavy proteinuria. Int Urol Nephrol. 2021 Jun;53(6):1197-1207. doi: 10.1007/s11255-020-02717-2. Epub 2021 Jan 2. PMID 33389459